CLINICAL TRIAL: NCT03288051
Title: Effects of Intraoperative, Goal-directed Crystalloid vs. Colloid Fluid Resuscitation on Microcirculation in Free Flap Reconstruction of Intraoral Tumours.
Brief Title: Effects of Intraoperative, Goal-directed Crystalloid vs. Colloid Fluid Resuscitation on Free Flaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Szeged University (Other)
Collaborators: Department of Oral and Maxillofacial Surgery, University of Szeged (Unknown); Institute of Surgical Research, University of Szeged (Unknown)
Responsible Party: Principal Investigator, Zsolt Molnár, MD, PhD, DEAA, head of department, Szeged University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Free Flap Microcirculation
Record Dates: First submitted 2017-08-29; First posted 2017-09-19 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Optimal Tissue Perfusion
MeSH Terms: interventions — Norepinephrine; Dobutamine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crystalloid group (Active Comparator)
  Interventions: Other: Fluid management; Drug: Norepinephrine; Drug: Dobutamine
- Colloid group (Active Comparator)
  Interventions: Other: Fluid management; Drug: Norepinephrine; Drug: Dobutamine

INTERVENTIONS:
Other: Fluid management — Primary fluid admission: 1 mL/bodyweight kg/ hour crystalloid. If Pulse pressure variation is lower than 10%; 250 mL/15 min of colloid or crystalloid is administered depending on randomization.
Drug: Norepinephrine — Norepinephrine is administered if Mean arterial pressure drops below 65 mmHg. Mean arterial pressure must be maintained above 65 mmHg. Norepinephrine is titrated accordingly.
Drug: Dobutamine — Dobutamine is administered if Cardiac index drops below 2.5 L/min/m2. Cardiac index must be maintained above 2.5 L/min/m2. Dobutamine is titrated accordingly.

SUMMARY:
Maintaining satisfactory tissue perfusion is an essential of success during reconstructive free flap surgery following malign oral cavity tumours. Intra- and postoperative goal-directed fluid therapy is an appropriate tool for that. Continuous cardiac output monitoring based fluid loading (complemented with vasopressor and/or inotropes if necessary) might be superior to conventional, central venous and arterial pressure monitoring in terms of morbidity, complications, optimal fluid balance and days spent in hospital. However, there is no data describing the effects of goal-directed fluid therapy (crystalloid or colloid) on microcirculation of free flaps implanted in the oral cavity during the post-operative period. The aim of this study is to observe the effects of continuous macrohaemodynamic monitoring based, goal-directed fluid therapy on microcirculation of forearm flaps during the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Tumour location: intraoral
* Free flap type: radial forearm
* Signed informed concent form

Exclusion Criteria:

* Vulnerable subject as defined in International Standards Organization 14155:2011
* End stage oral cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04-28 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
Changes of Pulse pressure variation during the operation and the post-operative 24 hours | 24 hours
Assesment of free falp microcirculation by laser dopler flowmetry method. | 24 hours
Total need of Norepinephrine and Dobutamine during surgery and the post-operative 24 hours. | 24 hours
Changes of Cardiac Index during the operation and the post-operative 24 hours. | 24 hours
Mean arterial pressure during the operation and the post-operative 24 hours. | 24 hours

SECONDARY OUTCOMES:
Length of Intensive Care Unit stay | 24 hours
Number of surgical or non-surgical complications. | 24 hours
Length of Hospital stay | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Intensive Therapy, Szeged, Csongrád megye, Hungary

REFERENCES:
- [Background] Salzwedel C, Puig J, Carstens A, Bein B, Molnar Z, Kiss K, Hussain A, Belda J, Kirov MY, Sakka SG, Reuter DA. Perioperative goal-directed hemodynamic therapy based on radial arterial pulse pressure variation and continuous cardiac index trending reduces postoperative complications after major abdominal surgery: a multi-center, prospective, randomized study. Crit Care. 2013 Sep 8;17(5):R191. doi: 10.1186/cc12885. PMID 24010849
- [Background] Holzle F, Rau A, Loeffelbein DJ, Mucke T, Kesting MR, Wolff KD. Results of monitoring fasciocutaneous, myocutaneous, osteocutaneous and perforator flaps: 4-year experience with 166 cases. Int J Oral Maxillofac Surg. 2010 Jan;39(1):21-8. doi: 10.1016/j.ijom.2009.10.012. Epub 2009 Nov 26. PMID 19944567
- [Background] Cecconi M, Hofer C, Teboul JL, Pettila V, Wilkman E, Molnar Z, Della Rocca G, Aldecoa C, Artigas A, Jog S, Sander M, Spies C, Lefrant JY, De Backer D; FENICE Investigators; ESICM Trial Group. Fluid challenges in intensive care: the FENICE study: A global inception cohort study. Intensive Care Med. 2015 Sep;41(9):1529-37. doi: 10.1007/s00134-015-3850-x. Epub 2015 Jul 11. PMID 26162676
- [Derived] Laszlo I, Janovszky A, Lovas A, Vargan V, Oveges N, Tanczos T, Mikor A, Trasy D, Loderer Z, Piffko J, Szabo A, Molnar Z. Effects of goal-directed crystalloid vs. colloid fluid therapy on microcirculation during free flap surgery: A randomised clinical trial. Eur J Anaesthesiol. 2019 Aug;36(8):592-604. doi: 10.1097/EJA.0000000000001024. PMID 31157652